CLINICAL TRIAL: NCT03015571
Title: Influence of Routine Use of Narrow Band Imaging on Heterotopic Gastric Mucosa of the Proximal Esophagus Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomasz Romańczyk (Other)
Responsible Party: Sponsor-Investigator, Tomasz Romańczyk, Principal Investigator Tomasz Romańczyk MD, PhD, H-T. Centrum Medyczne Sp. z o.o. sp. k
Organization: H-T. Centrum Medyczne Sp. z o.o. sp. k (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HT-001
Record Dates: First submitted 2016-12-29; First posted 2017-01-10 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Heterotopic Gastric Mucosa of the Proximal Esophagus
Keywords: heterotopic gastric mucosa; cervical inlet patch; narrow band imaging; endoscopy
MeSH Terms: interventions — Narrow Band Imaging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- NBI (Experimental): Use of Narrow Band Imaging with regular care of cervical inlet patches detection.
  Interventions: Device: Esophagus inspection in Narrow Band imaging.
- WL (Placebo Comparator): Use of High Definition White Light (WL) with regular care of cervical inlet patches detection.
  Interventions: Device: Standard High definition endoscopy.
- NBI increased care (Experimental): Use of Narrow Band Imaging with increased care of cervical inlet patches detection.
  Interventions: Device: Esophagus inspection in Narrow Band imaging and increased care.
- WL increased care (Placebo Comparator): Use of High Definition White Light (WL) with increased care of cervical inlet patches detection.
  Interventions: Device: Standard High definition endoscopy and increased care.

INTERVENTIONS:
Device: Esophagus inspection in Narrow Band imaging. — During the endoscope withdrawal after cardia examination NBI will be used for esophagus inspection.
  Arms: NBI
Device: Standard High definition endoscopy. — Whole procedure will be performed in standard High definition endoscopy.
  Arms: WL
Device: Esophagus inspection in Narrow Band imaging and increased care. — During the endoscope withdrawal after cardia examination NBI will be used for esophagus inspection and with increased care of cervical inlet patches detection.
  Arms: NBI increased care
Device: Standard High definition endoscopy and increased care. — Whole procedure will be performed in standard High definition endoscopy with increased care of cervical inlet patches detection.
  Arms: WL increased care

SUMMARY:
The aim of the study is to determine whether Narrow Band Imaging(NBI) should be routinely used during esophagus inspection at diagnostic gastroscopy.

DETAILED DESCRIPTION:
Heterotopic gastric mucosa, also called inlet patch, is area of ectopic gastric mucosa with common location at proximal part of esophagus. Because of the location, lesions are likely to be missed during routine gastroscopy. The clinical significance of inlet patches remains unknown, however they may be symptomatic and may cause morphologic changes such as strictures, ulcers, webs, stenoses or even adenocarcinomas. Moreover inlet patches may be correlated with reflux symptoms up to 73,1%. Several studies were conducted to determine whether NBI improves detection of cervical inlet patches, some of them were also prospective studies, however no randomized study was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Referral for diagnostic gastroscopy
* Ability to undergo diagnostic gastroscopy
* Provided written informed consent

Exclusion Criteria:

* Age <18
* Prisoners
* Pregnancy
* Gastroscopy with treatment procedure
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
Detection of heterotopic gastric mucosa in the proximal esophagus | Day 1

SECONDARY OUTCOMES:
Total and esophagus inspection time | Day 1
Detection of other upper gastrointestinal lesions | Day 1
Correlation of throat and esophageal reflux symptoms with cervical inlet patches | Day 1
Rate of cervical inlet patches verified with NBI in endoscopies performed in standard white light endoscopy | Day 1
Correlation of subject's subjective purpose of gastroscopy and cervical inlet patch occurrence | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- H-T.Centrum Medyczne Sp. z o.o. Sp. K., Tychy, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] von Rahden BH, Stein HJ, Becker K, Liebermann-Meffert D, Siewert JR. Heterotopic gastric mucosa of the esophagus: literature-review and proposal of a clinicopathologic classification. Am J Gastroenterol. 2004 Mar;99(3):543-51. doi: 10.1111/j.1572-0241.2004.04082.x. PMID 15056100
- [Background] Maconi G, Pace F, Vago L, Carsana L, Bargiggia S, Bianchi Porro G. Prevalence and clinical features of heterotopic gastric mucosa in the upper oesophagus (inlet patch). Eur J Gastroenterol Hepatol. 2000 Jul;12(7):745-9. doi: 10.1097/00042737-200012070-00005. PMID 10929900
- [Background] Chong VH. Clinical significance of heterotopic gastric mucosal patch of the proximal esophagus. World J Gastroenterol. 2013 Jan 21;19(3):331-8. doi: 10.3748/wjg.v19.i3.331. PMID 23372354
- [Background] Chong VH, Jalihal A. Heterotopic gastric mucosal patch of the esophagus is associated with higher prevalence of laryngopharyngeal reflux symptoms. Eur Arch Otorhinolaryngol. 2010 Nov;267(11):1793-9. doi: 10.1007/s00405-010-1259-2. Epub 2010 May 1. PMID 20437050
- [Background] Al-Mammari S, Selvarajah U, East JE, Bailey AA, Braden B. Narrow band imaging facilitates detection of inlet patches in the cervical oesophagus. Dig Liver Dis. 2014 Aug;46(8):716-9. doi: 10.1016/j.dld.2014.05.001. Epub 2014 Jun 2. PMID 24890619
- [Background] Cheng CL, Lin CH, Liu NJ, Tang JH, Kuo YL, Tsui YN. Endoscopic diagnosis of cervical esophageal heterotopic gastric mucosa with conventional and narrow-band images. World J Gastroenterol. 2014 Jan 7;20(1):242-9. doi: 10.3748/wjg.v20.i1.242. PMID 24415878
- [Background] Chung CS, Lin CK, Liang CC, Hsu WF, Lee TH. Intentional examination of esophagus by narrow-band imaging endoscopy increases detection rate of cervical inlet patch. Dis Esophagus. 2015 Oct;28(7):666-72. doi: 10.1111/dote.12252. Epub 2014 Jul 24. PMID 25059461
- [Background] Vesper I, Schmiegel W, Brechmann T. Equal detection rate of cervical heterotopic gastric mucosa in standard white light, high definition and narrow band imaging endoscopy. Z Gastroenterol. 2015 Nov;53(11):1247-54. doi: 10.1055/s-0041-104226. Epub 2015 Nov 12. PMID 26562398
- [Background] Azar C, Jamali F, Tamim H, Abdul-Baki H, Soweid A. Prevalence of endoscopically identified heterotopic gastric mucosa in the proximal esophagus: endoscopist dependent? J Clin Gastroenterol. 2007 May-Jun;41(5):468-71. doi: 10.1097/01.mcg.0000225519.59030.8d. PMID 17450028
- [Derived] Romanczyk M, Budzyn K, Romanczyk T, Lesinska M, Koziej M, Hartleb M, Waluga M. Heterotopic Gastric Mucosa in the Proximal Esophagus: Prospective Study and Systematic Review on Relationships with Endoscopic Findings and Clinical Data. Dysphagia. 2023 Apr;38(2):629-640. doi: 10.1007/s00455-022-10492-8. Epub 2022 Jul 9. PMID 35809096
- [Derived] Romanczyk M, Romanczyk T, Lesinska M, Romanczyk A, Hartleb M, Waluga M. Influence of narrow-band imaging (NBI) and enhanced operator's attention during esophagus inspection on cervical inlet patches detection. Adv Med Sci. 2021 Mar;66(1):170-175. doi: 10.1016/j.advms.2021.02.002. Epub 2021 Feb 25. PMID 33640715
- See also: Incidence of Heterotopic Gastric Mucosa in the Upper Esophagus in First Time Narrow Banding Image Endoscopy. — http://www.giejournal.org/article/S0016-5107(10)01071-0/fulltext